CLINICAL TRIAL: NCT05510323
Title: Efficacy and Safety of Immunosuppressive Therapy for IgA Nephropathy With Stage 3 or 4 Chronic Kidney Disease
Brief Title: Efficacy of Immunosuppressive Therapy for IgA Nephropathy With Stage 3 or 4 CKD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Shiren sun, Chief, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20222108-F-1
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Glomerulonephritis, IGA
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Prednisolone; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CS (Active Comparator): low-dose corticosteroids monotherapy
  Interventions: Drug: Prednisolone
- CS+CTX (Active Comparator): low-dose corticosteroids combined with cyclophosphamide
  Interventions: Drug: Prednisolone plus Cyclophosphamide

INTERVENTIONS:
Drug: Prednisolone — RAS blockade as much as tolerated or allowed
  Arms: CS
Drug: Prednisolone plus Cyclophosphamide — RAS blockade as much as tolerated or allowed
  Arms: CS+CTX

SUMMARY:
The purpose of this clinical trial is to evaluate the long-term efficacy and safety of low-dose oral corticosteroids combined with cyclophosphamide therapy and low-dose corticosteroids monotherapy, on a background of maximal RAS inhibitor therapy, for IgA nephropathy with stage 3 or 4 chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven IgA nephropathy;
* Proteinuria ≥1.0g/day while receiving maximum tolerated dose of RAS blockade;
* Estimated glomerular filtration rate 15-60 ml/min/1.73/m2.

Exclusion Criteria:

* Indication or contraindication for immunosuppressive therapy with corticosteroids
* Use of corticosteroids and other immunosuppressive drugs within the last 1 year
* Current unstable kidney function for other reasons
* Under 18 years old
* Patients with secondary IgAN
* Patients who are unlikely to comply with the study protocol in the view of the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Combined event | up to 6 years
  40% decrease in eGFR, ESRD or death due to kidney disease

SECONDARY OUTCOMES:
Proteinuria remission at 6, 12 months and total follow-up period | up to 6 years
  Proteinuria remission
Hematuria remission at 6, 12 months and total follow-up period | up to 6 years
  Hematuria remission
The composite of 30% decrease in eGFR, ESRD and all cause death | up to 6 years
The composite of 40% decrease in eGFR, ESRD and all cause death | up to 6 years
The composite of 50% decrease in eGFR, ESRD and all cause death | up to 6 years
Annual eGFR decline rate | up to 6 years
30% decrease in eGFR | up to 6 years
40% decrease in eGFR | up to 6 years
50% decrease in eGFR | up to 6 years
ESRD | up to 6 years
All cause death | up to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- AFMMU, Xi'an, China